CLINICAL TRIAL: NCT01715233
Title: A Phase II Study Investigating CHFR Methylation Status As A Biomarker For Taxane Sensitivity Using Modified Docetaxel, Cisplatin and 5 Fluorouracil In Patients With Metastatic Esophageal, Gastroesophageal And Gastric Cancer.
Brief Title: Phase II Study Using CHFR Methylation Status in Patients With Metastatic Esophageal, Gastroesophageal, Gastric Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1248; NA_00073720 (Other: JHM IRB)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Esophageal Cancer; Gastroesophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Docetaxel; Leucovorin; Fluorouracil; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metastatic Esophageal, Gastroesophageal & Gastric Cancer (Experimental): Participants receive Modified Docetaxel 40mg/m2, Leucovorin 400mg/m2 and Fluorouracil 400mg/m2 on day 1, Fluorouracil 1000mg/m2 per day on days 1 and 2 and Cisplatin 40mg/m2 (or Carboplatin) on day 3 in Patients With Metastatic Esophageal, Gastroesophageal And Gastric Cancer.
  Interventions: Drug: Docetaxel; Drug: Leucovorin; Drug: Fluorouracil; Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel — Modified Docetaxel 40mg/m2 on Day 1
  Other Names: Modified DCF
Drug: Leucovorin — Leucovorin 400mg/m2 on Day 1
Drug: Fluorouracil — Fluorouracil 400mg/m2 on Day 1 Fluorouracil 1000mg/m2/day on Days 1 and 2
  Other Names: FU
Drug: Cisplatin — Cisplatin (or Carboplatin) 40mg/m2 on Day 3
  Other Names: Carboplatin

SUMMARY:
To estimate and compare the response rates in patients treated with mDCF based on methylation status of CHFR.

DETAILED DESCRIPTION:
To estimate and compare the response rates in patients treated with mDCF based on methylation status of CHFR. The overall response rates in the un-methylated and methylated patient groups will be reported with a exact 95% binomial confidence interval. A chi-square test will be used for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic disease of the esophagus, gastroesophageal junction or stomach. Patients with locally recurrent disease who are not deemed eligible for radiation are also permitted.
* Histological, cytologic or radiographic documentation of metastatic adenocarcinoma or squamous cell carcinoma of the esophagus, gastroesophageal junction or stomach. Radiologic, endoscopic, histologic or cytologic evidence of locally recurrent disease is also permitted.
* Patients must be untreated with chemotherapy for metastatic or locally recurrent disease. Prior radiation therapy is permitted.
* Patients must have measurable disease as per RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Age >18 years and ≤ 80 years.
* ECOG performance status <2 (Karnofsky >60%, see Appendix A).
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function.
* Patients must not have any of the following conditions:
* Recent major surgery, hormonal therapy (other than replacement) or chemotherapy, within 4 weeks prior to entering the study or those who have not recovered from the adverse events of treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the chemotherapy on this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the chemotherapy used in the study.
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St John's Wort; these drugs induce CYP3A and may decrease levels of taxanes. 5-FU is a strong CYP2C9 inducer, and concomitant use with carvedilol, celecoxib, fosphenytoin, fluoxetine, phenytoin, warfarin and other CYP2C9 substrates should be used with caution.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because chemotherapy has the potential for teratogenic or abortifacient effects.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with chemotherapeutic agents. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronan J Kelly, MD, MBA, Principal Investigator — SKCCC at Johns Hopkins
Locations (1):
- SKCCC at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 subjects were screen failures.
Period: Overall Study
Arm/Group | Metastatic Esophageal, Gastroesophageal & Gastric Cancer
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metastatic Esophageal, Gastroesophageal & Gastric Cancer
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Number of participants treated with mDCF with progressive disease (PD), stable disease (SD), partial response (PR), non-complete response and non-progressive disease (non-CR/non-PD), and partial response with progressive disease clinically (PR/PD) as defined by RECIST criteria. Response is compared based on CHFR-methylation status.
Time Frame: 4 months
Population: Response could not be assessed in 2/21 participants since imaging was not evaluable, therefore RECIST reads could not be obtained.
Measure: Count of Participants; unit: Participants
Groups:
- Metastatic Esophageal, Gastroesophageal & Gastric Cancer.: Participants receive Modified Docetaxel 40mg/m2, Leucovorin 400mg/m2 and Fluorouracil 400mg/m2 on day 1, Fluorouracil 1000mg/m2 per day on days 1 and 2 and Cisplatin 40mg/m2 (or Carboplatin) on day 3 in Patients With Metastatic Esophageal, Gastroesophageal And Gastric Cancer.
  Docetaxel: Modified Docetaxel 40mg/m2 on Day 1 Leucovorin: Leucovorin 400mg/m2 on Day 1 Fluorouracil: Fluorouracil 400mg/m2 on Day 1 Fluorouracil 1000mg/m2/day on Days 1 and 2 Cisplatin: Cisplatin (or Carboplatin) 40mg/m2 on Day 3
Arm/Group | Metastatic Esophageal, Gastroesophageal & Gastric Cancer.
Number analyzed (Participants) | 19
Participants
  CHFR-methylated: number analyzed (Participants) | 6
  CHFR-methylated: PD | 3
  CHFR-methylated: SD | 0
  CHFR-methylated: PR | 2
  CHFR-methylated: non-CR/non-PD | 0
  CHFR-methylated: PR/PD | 1
  CHFR-unmethylated: number analyzed (Participants) | 12
  CHFR-unmethylated: PD | 3
  CHFR-unmethylated: SD | 3
  CHFR-unmethylated: PR | 5
  CHFR-unmethylated: non-CR/non-PD | 1
  CHFR-unmethylated: PR/PD | 0
  Unknown methylation status: number analyzed (Participants) | 1
  Unknown methylation status: PD | 0
  Unknown methylation status: SD | 0
  Unknown methylation status: PR | 1
  Unknown methylation status: non-CR/non-PD | 0
  Unknown methylation status: PR/PD | 0

2. Secondary Outcome: CHFR Methylation Status
Description: Number of participants with advanced esophagogastric cancer that are CHFR-methylated or unmethylated at baseline.
Time Frame: Baseline
Population: Only 18/21 participants had evaluable data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Metastatic Esophageal, Gastroesophageal & Gastric Cancer.
Number analyzed (Participants) | 18
Participants
  CHFR-methylated | 6
  CHFR-unmethylated | 12

3. Secondary Outcome: Overall Survival
Description: Number of participants alive at 2 years.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Groups:
- Metastatic Esophageal, Gastroesophageal And Gastric Cancer.: Participants receive Modified Docetaxel 40mg/m2, Leucovorin 400mg/m2 and Fluorouracil 400mg/m2 on day 1, Fluorouracil 1000mg/m2 per day on days 1 and 2 and Cisplatin 40mg/m2 (or Carboplatin) on day 3 in Patients With Metastatic Esophageal, Gastroesophageal And Gastric Cancer.
  Docetaxel: Modified Docetaxel 40mg/m2 on Day 1 Leucovorin: Leucovorin 400mg/m2 on Day 1 Fluorouracil: Fluorouracil 400mg/m2 on Day 1 Fluorouracil 1000mg/m2/day on Days 1 and 2 Cisplatin: Cisplatin (or Carboplatin) 40mg/m2 on Day 3
Arm/Group | Metastatic Esophageal, Gastroesophageal And Gastric Cancer.
Number analyzed (Participants) | 21
Participants | 2

ADVERSE EVENTS:
Time Frame: AEs assessed during each study visit for up to 1 year; All-Cause Mortality was assessed for up to 2 years.
Description: Only Grades 3 and 4 adverse events were collected for all patients.
Groups:
- Metastatic Esophageal, Gastroesophageal & Gastric Cancer: Patients received modified Docetaxel 40mg/m2, Leucovorin 400mg/m2 and Fluorouracil 400mg/m2 on day 1, Fluorouracil 1000mg/m2 per day on days 1 and 2 and Cisplatin 40mg/m2 (or Carboplatin) on day 3 in Patients With Metastatic Esophageal, Gastroesophageal And Gastric Cancer.
  Docetaxel: Modified Docetaxel 40mg/m2 on Day 1
  Leucovorin: Leucovorin 400mg/m2 on Day 1
  Fluorouracil: Fluorouracil 400mg/m2 on Day 1 Fluorouracil 1000mg/m2/day on Days 1 and 2
  Cisplatin: Cisplatin (or Carboplatin) 40mg/m2 on Day 3
Arm/Group | Metastatic Esophageal, Gastroesophageal & Gastric Cancer
All-Cause Mortality (participants affected / at risk) | 19/21
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic Esophageal, Gastroesophageal & Gastric Cancer (N=21)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytopenia (Blood and lymphatic system disorders) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic Esophageal, Gastroesophageal & Gastric Cancer (N=21)
Hospitalization due to leg pain (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytopenia (Blood and lymphatic system disorders) | 5 (9)
Dehydration (Gastrointestinal disorders) | 1 (1)
Fainting (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hypotensive (Cardiac disorders) | 1 (1)
Increased INR (Vascular disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 3 (9)
Lymphopenia (Blood and lymphatic system disorders) | 5 (7)
Neutropenia (Blood and lymphatic system disorders) | 11 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No